CLINICAL TRIAL: NCT02432781
Title: Effect of Preoperative Oral Carbohydrates on Postoperative Nausea and Vomiting and Quality of Recovery in DM Patients Undergoing Total Knee Arthroplasty
Brief Title: Oral Carbohydrate in DM Patients Undergoing Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Assistant professor, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4-2015-0151
Record Dates: First submitted 2015-04-23; First posted 2015-05-04 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbohydrate group (Experimental): Carbohydrate-rich drink 400 mL 3 h before surgery
  Interventions: Dietary Supplement: Carbohydrate-rich drink
- Control group (Active Comparator): 10% dextrose solution mixed with insulin 16 unit 100 mL/h
  Interventions: Dietary Supplement: 10% dextrose solution mixed with insulin 16 unit 100 mL/h

INTERVENTIONS:
Dietary Supplement: Carbohydrate-rich drink
  Arms: Carbohydrate group
Dietary Supplement: 10% dextrose solution mixed with insulin 16 unit 100 mL/h
  Arms: Control group

SUMMARY:
The primary purpose of this study is to investigate the effects of carbohydrate-rich drink on postoperative nausea and vomiting in diabetic patients undergoing total knee arthroplasty. The secondary purpose is to investigate the effects of carbohydrate-rich drink on quality of recovery and inflammation in diabetic patients after total knee arthroplasty.

DETAILED DESCRIPTION:
Carbohydrate-rich drink has been proved to neither delay gastric emptying nor affect gastric acidity and is therefore considered safe to use in elective surgical patients without risk factors for pulmonary aspiration. It reduced postoperative nausea and vomiting and improved sense of well-being after surgery. Moreover, carbohydrate-rich drink was not found to be affected by delayed gastric emptying in patients with uncomplicated type 2 diabetes. Therefore, carbohydrate drink may be safely administered 3 h before anesthesia without risk of hyperglycemia or aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 DM patients undergoing elective total knee arthroplasty

Exclusion Criteria:

* Contraindication to regional anesthesia
* Patients whose operation is scheduled to start after 9:00 am
* Dementia or cognitive dysfunction
* HbA1c > 8%
* Gastroesophageal reflux disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting | 24 hours

SECONDARY OUTCOMES:
Score of quality of recovery | 24 hours
  Quality of recovery is determined by a 40-item quality-of-recovery questionnaire
Degree of inflammation | 24 hours
  Degree of inflammation is determined by white blood cell count, neutrophil count, and C-reactive protein

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Shin S, Choi YS, Shin H, Yang IH, Park KK, Kwon HM, Kang B, Kim SY. Preoperative Carbohydrate Drinks Do Not Decrease Postoperative Nausea and Vomiting in Type 2 Diabetic Patients Undergoing Total Knee Arthroplasty-A Randomized Controlled Trial. J Am Acad Orthop Surg. 2021 Jan 1;29(1):35-43. doi: 10.5435/JAAOS-D-20-00089. PMID 32433428